CLINICAL TRIAL: NCT02349295
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled 24-Week Study Followed by Long Term Evaluation of Efficacy and Safety of Ixekizumab (LY2439821) in Biologic Disease-Modifying Antirheumatic Drug-Experienced Patients With Active Psoriatic Arthritis
Brief Title: A Study of Ixekizumab (LY2439821) in Participants With Active Psoriatic Arthritis
Acronym: SPIRIT-P2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14310; I1F-MC-RHBE (Other: Eli Lilly and Company); 2011-002328-42 (EudraCT Number)
Record Dates: First submitted 2014-10-10; First posted 2015-01-28 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2019-09-01

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ixekizumab 80 milligram (mg) every 2 Weeks (Q2W) (Experimental): Blinded Treatment Period (Week(wk) 0-24): Participants (pts) received a starting dose of 160 mg of ixekizumab (ixe) given as 2 subcutaneous (SC) injections at Wk 0 followed by 1 SC injection of 80 mg of ixe Q2W given on Wks 2,4,6,8,10,12,14,16,18,20,22, and 24.Week 16 inadequate responders (IR) from the placebo treatment group who were re-randomized (1:1) to ixe 80 mg Q2W and IR from ixekizumab 80 mg Q2W who continued on ixekizumab 80 mg Q2W. Pts receive rescue therapy while receiving ixekizumab given as 1 injection of 80 mg Q2W given on Wks 16,18,20,22,24. Extension Period (Wk24-156):Pts who were randomized to ixe 80 mg Q2W at week 0 and continued on ixe 80 mg Q2W during the Extension Period. Pts who received ixekizumab 80 mg Q2W,who were either completed the study or discontinued the study early entered the post-treatment follow-up period (12-24 weeks).
  Interventions: Drug: Placebo; Drug: Ixekizumab 80 mg Q2W
- Ixekizumab 80 mg Q4W (Experimental): Blinded Treatment Period (Week 0-24): Participants (pts) received a starting dose of 160 mg of ixekizumab (ixe) given as 2 subcutaneous (SC) injections at Wk 0 followed by 1 SC injection of 80 mg of ixe Q4W given on Wks 4, 8 and 12 alternating with placebo for ixe injections Q4W given on Wks 2,6,10,14,18, and 22.Week 16 inadequate responders (IR) from the placebo treatment group who were re-randomized (1:1) to ixe 80 mg Q4W and IR from ixekizumab 80 mg Q4W who continued on ixekizumab 80 mg Q4W. Pts receive rescue therapy while receiving ixekizumab given as 1 injection of 80 mg Q4W given on Wks 16 and 20 alternating with placebo for ixe injections Q4W given on Wks 18 and 22.Extension Period (Wk24-156):Pts who were randomized to ixe 80 mg Q4W at week 0 and continued on ixe 80 mg Q4W during the Extension Period.Pts who received ixekizumab 80 mg Q4W,who were either completed the study or discontinued the study early entered the post-treatment follow-up period (12-24 weeks).
  Interventions: Drug: Placebo; Drug: Ixekizumab 80 mg Q4W
- Placebo (Placebo Comparator): Blinded Treatment Period (Wk 0-24): Pts received placebo for Ixe as 2 SC injections followed by 1 SC injection Q2W given on Wks 2,4,6,8,10,12,14,16,18,20,22 and 24. Pts initially randomized to placebo treatment group in the double blind treatment period,flagged as IR at Wk 16,re-randomized to ixe 80 mg Q2W/Q4W for the remainder of the current period and following period. Extended Treatment Period (Wk 24-156): Pts who were randomized to placebo at Week 0 then randomized to ixekizumab 80 mg Q2W/Q4W during the Extension Period.Pts who remained on placebo at the completion of the double blind treatment period received the first dose of ixe (160 mg starting dose) at Wk 24.Pts who were IRs at Wk 16 and were re-randomized to ixe at Wk 16 received the first dose of ixe (160 mg starting dose) at Wk 16. Pts who received placebo,who were either completed the study or discontinued the study early entered the post-treatment follow-up period (12-24 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Administered SC
Drug: Ixekizumab 80 mg Q4W — Administered SC
  Other Names: LY2439821
  Arms: Ixekizumab 80 mg Q4W
Drug: Ixekizumab 80 mg Q2W — Administered SC
  Other Names: LY2439821
  Arms: Ixekizumab 80 milligram (mg) every 2 Weeks (Q2W)

SUMMARY:
The main purpose of this study is to evaluate how effective and safe the study drug known as ixekizumab is in participants with active psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Presents with established diagnosis of active psoriatic arthritis (PsA) for at least 6 months, and currently meets Classification for Psoriatic Arthritis (CASPAR) criteria
* Active PsA defined as the presence of at least 3 tender and at least 3 swollen joints
* Presence of active psoriatic skin lesion or a history of plaque psoriasis (Ps)
* Men must agree to use a reliable method of birth control or remain abstinent during the study
* Women must agree to use reliable birth control or remain abstinent during the study and for at least 12 weeks after stopping treatment
* Have been treated with 1 or more conventional disease-modifying antirheumatic drugs (cDMARDs)
* Have had prior treatment with at least 1 and not more than 2 tumor necrosis factor (TNF) inhibitors. The participant must have discontinued at least 1 TNF inhibitor due to either an inadequate response (based on a minimum of 12 weeks on therapy) or documented intolerance.

Exclusion Criteria:

* Current use of biologic agents for treatment of Ps or PsA
* Inadequate response to greater than 2 biologic DMARDs
* Current use of more than one cDMARDs
* Diagnosis of active inflammatory arthritic syndromes or spondyloarthropathies other than PsA
* Have received treatment with interleukin (IL) -17 or IL12/23 targeted monoclonal antibody (MAb) therapy
* Serious disorder or illness other than psoriatic arthritis
* Serious infection within the last 3 months
* Breastfeeding or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2016-09-09 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (109):
- United States (59):
  - Rheumatology Associates PC, Birmingham, Alabama
  - Arizona Arthritis & Rheumatology Research, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Research, Phoenix, Arizona
  - Little Rock Diagnostic Clinic, Little Rock, Arkansas
  - University of California - San Diego, La Jolla, California
  - Purushotham & Akther Kotha MD Inc, La Mesa, California
  - Stanford University Hospital, Palo Alto, California
  - East Bay Rheumatology Medical Group, San Leandro, California
  - Office: Dr Robin K Dore, Tustin, California
  - Rheumatology Associates of South Florida, Boca Raton, Florida
  - Jeffrey Alper MD Research, Naples, Florida
  - Arthritis & Osteoporosis Treatment Center, PA, Orange Park, Florida
  - Florida Medical Clinic PA, Zephyrhills, Florida
  - Diagnostic Rheumatology and Research, Indianapolis, Indiana
  - Physicians Clinic of Iowa, Cedar Rapids, Iowa
  - Heartland Research Associates, Wichita, Kansas
  - Bluegrass Community Research. Inc, Lexington, Kentucky
  - Johns Hopkins Arthritis Center, Baltimore, Maryland
  - Klein and Associates MD, PA, Cumberland, Maryland
  - Klein and Associates MD, PA, Hagerstown, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beals Institute PC, Lansing, Michigan
  - North MS Medical Clinics, Inc., Tupelo, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Glacier View Research Institute, Kalispell, Montana
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - New Jersey Physicians, Clifton, New Jersey
  - Atlantic Coastal Research, Toms River, New Jersey
  - Arthritis, Rheumatic & Back Disease Associates, Voorhees Township, New Jersey
  - Albuquerque Rehabilitation & Rheumatology, PC, Albuquerque, New Mexico
  - The Center for Rheumatology, Albany, New York
  - Weill Cornell Medical College, Brooklyn, New York
  - Allergy Asthma Immunology of Rochester, AAIR Research Ctr, Rochester, New York
  - Rheumatology Associates of Long Island, Smithtown, New York
  - Arthritis and Osteoporosis Consultants of the Carolinas, Charlotte, North Carolina
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - STAT Research, Dayton, Ohio
  - Health Research Institute, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - PMA Medical Specialists, LLC, Limerick, Pennsylvania
  - Clinical Research Center of Reading, LLC, Wyomissing, Pennsylvania
  - Pennsylvania Regional Center for Arthritis & Osteoarthritis, Wyomissing, Pennsylvania
  - Methodist Healthcare, Memphis, Tennessee
  - Ramesh C. Gupta MD, Memphis, Tennessee
  - Austin Rheumatology Research PA, Austin, Texas
  - Austin Regional Clinic, Austin, Texas
  - Arthritis Care & Diagnostic Center P.A., Dallas, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Houston Institute for Clinical Research, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Accurate Clinical Research, League City, Texas
  - Arthritis & Osteoporosis Associates LLP, Lubbock, Texas
  - Kadlec Clinic Rheumatology, Kennewick, Washington
  - Swedish Medical Center, Seattle, Washington
  - Arthritis Northwest PLLC, Spokane, Washington
  - Rheumatology and Immunotherapy Center, Franklin, Wisconsin
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Coast Joint Care, Maroochydore, Queensland
  - Emeritus Research, Camberwell, Victoria
- Czechia (3):
  - CCBR Czech Prague, s.r.o., Prague
  - MEDICAL PLUS, s.r.o., Uherské Hradiště
  - PV-MEDICAL s.r.o. Revmatologicka ambulance, Zlín
- France (6):
  - Hôpital Trousseau, CHRU de Tours, Chambray-lès-Tours
  - CHU de Montpellier-Hopital Arnaud de Villeneuve, Montpellier
  - Chru De Nantes Hotel-Dieu, Nantes
  - Hopital Cochin, Paris
  - Hopital Purpan, Toulouse
  - CHU Brabois, Vandœuvre-lès-Nancy
- Germany (10):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt am Main, Hesse
  - Rheumazentrum Ruhrgebiet, Herne, North Rhine-Westphalia
  - Krankenhaus Dresden-Friedrichstadt Städtisches Klinikum, Dresden, Saxony
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universität Leipzig - Universitätsklinikum, Leipzig, Saxony
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Charité Universitätsmedizin Berlin, Berlin
  - HRF Hamburger Rheuma Forschungszentrum, Hamburg
- Italy (2):
  - Istituto Ortopedico Gaetano Pini, Milan
  - Azienda Ospedaliera - Universitaria Pisana, Pisa
- Poland (5):
  - Malopolskie Centrum Medyczne S.C., Krakow
  - Medica pro Familia Sp z o.o. S.K.A, Krakow
  - AI Centrum Medyczne, Poznan
  - Medica pro Familia Sp z o.o. S.K.A, Warsaw
  - Rheuma Medicus Zakład Opieki Zdrowotnej, Warsaw
- Spain (8):
  - Hospital Infanta Luisa, Seville, Andalusia
  - Centro de Salud Mental Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Marques De Valdecilla, Santander, Cantabria
  - Hospital De Fuenlabrada, Fuenlabrada, Madrid
  - Hospital De Basurto, Bilbao, Vizcaya
  - Complexo Hospitalario Universitario A Coruña, CHUAC, A Coruña
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Nuestra Señora de Valme, Seville
- Taiwan (7):
  - Chi-Mei Hospital, Liouying, Tainan, Yongkang Dist
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung City (r.o.c)
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan
- United Kingdom (6):
  - Basildon and Thurrock University Hospital, Basildon, Essex
  - King George Hospital, Goodmayes, Essex
  - Princess Alexandra Hospital, Harlow, Essex
  - Whipps Cross University Hospital, London, Surrey
  - New Cross Hospital, Wolverhampton, West Midlands
  - Chapel Allerton Hospital, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and european union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Kristensen LE, McGonagle D, Rudwaleit M, Kameda H, Wurtzen PA, Ngantcha M, Holzkamper T, Smolen J. Synergistic Improvements in Synovitis, Enthesitis, and Patient-Reported Outcomes for Patients with Psoriatic Arthritis Treated with Ixekizumab in SPIRIT Trials. Rheumatol Ther. 2025 Apr;12(2):381-395. doi: 10.1007/s40744-025-00748-8. Epub 2025 Feb 27. PMID 40014255
- [Derived] Tillett W, Birt J, Vadhariya A, Ross S, Ngantcha M, Ng KJ. Filling the "GAP" in Real-World Assessment of Psoriatic Arthritis Disease Activity: Performance Characteristics of a Global/Pain Composite Endpoint. Rheumatol Ther. 2024 Oct;11(5):1101-1114. doi: 10.1007/s40744-024-00690-1. Epub 2024 Jul 2. PMID 38955921
- [Derived] Armstrong AW, Jaleel T, Merola JF, Gottlieb AB, Khattri S, Helt CC, Malatestinic WN, Ross SE, Ngantcha ME, de Vlam K. Ixekizumab Demonstrates Rapid and Consistent Efficacy for Patients with Psoriatic Arthritis, Regardless of Psoriasis Severity. Dermatol Ther (Heidelb). 2024 Jun;14(6):1615-1631. doi: 10.1007/s13555-024-01188-y. Epub 2024 May 30. PMID 38814433
- [Derived] Kirkham BW, Egeberg A, Behrens F, Pinter A, Merola JF, Holzkamper T, Gallo G, Ng KJ, Bolce R, Schuster C, Nash P, Puig L. A Comprehensive Review of Ixekizumab Efficacy in Nail Psoriasis from Clinical Trials for Moderate-to-Severe Psoriasis and Psoriatic Arthritis. Rheumatol Ther. 2023 Oct;10(5):1127-1146. doi: 10.1007/s40744-023-00553-1. Epub 2023 Jul 3. PMID 37400681
- [Derived] Eder L, Tony HP, Odhav S, Agirregoikoa EG, Korkosz M, Schwartzman S, Sprabery AT, Gellett AM, Park SY, Bertram CC, Ogdie A. Responses to Ixekizumab in Male and Female Patients with Psoriatic Arthritis: Results from Two Randomized, Phase 3 Clinical Trials. Rheumatol Ther. 2022 Jun;9(3):919-933. doi: 10.1007/s40744-022-00445-w. Epub 2022 Apr 9. PMID 35397092
- [Derived] Deodhar AA, Combe B, Accioly AP, Bolce R, Zhu D, Gellett AM, Sprabery AT, Burmester GR. Safety of ixekizumab in patients with psoriatic arthritis: data from four clinical trials with over 2000 patient-years of exposure. Ann Rheum Dis. 2022 Jul;81(7):944-950. doi: 10.1136/annrheumdis-2021-222027. Epub 2022 Apr 7. PMID 35393269
- [Derived] Combe B, Tsai TF, Huffstutter JE, Sprabery AT, Lin CY, Park SY, Kronbergs A, Hufford MM, Nash P. Ixekizumab, with or without concomitant methotrexate, improves signs and symptoms of PsA: week 52 results from Spirit-P1 and Spirit-P2 studies. Arthritis Res Ther. 2021 Jan 27;23(1):41. doi: 10.1186/s13075-020-02388-5. PMID 33499913
- [Derived] Orbai AM, Gratacos J, Turkiewicz A, Hall S, Dokoupilova E, Combe B, Nash P, Gallo G, Bertram CC, Gellett AM, Sprabery AT, Birt J, Macpherson L, Geneus VJ, Constantin A. Efficacy and Safety of Ixekizumab in Patients with Psoriatic Arthritis and Inadequate Response to TNF Inhibitors: 3-Year Follow-Up (SPIRIT-P2). Rheumatol Ther. 2021 Mar;8(1):199-217. doi: 10.1007/s40744-020-00261-0. Epub 2020 Dec 5. PMID 33278016
- [Derived] Schweikert B, Malmberg C, Nunez M, Dilla T, Sapin C, Hartz S. Cost-effectiveness analysis of ixekizumab versus secukinumab in patients with psoriatic arthritis and concomitant moderate-to-severe psoriasis in Spain. BMJ Open. 2020 Aug 13;10(8):e032552. doi: 10.1136/bmjopen-2019-032552. PMID 32792421
- [Derived] Combe B, Rahman P, Kameda H, Canete JD, Gallo G, Agada N, Xu W, Genovese MC. Safety results of ixekizumab with 1822.2 patient-years of exposure: an integrated analysis of 3 clinical trials in adult patients with psoriatic arthritis. Arthritis Res Ther. 2020 Jan 21;22(1):14. doi: 10.1186/s13075-020-2099-0. PMID 31964419
- [Derived] Tillett W, Lin CY, Zbrozek A, Sprabery AT, Birt J. A Threshold of Meaning for Work Disability Improvement in Psoriatic Arthritis Measured by the Work Productivity and Activity Impairment Questionnaire. Rheumatol Ther. 2019 Sep;6(3):379-391. doi: 10.1007/s40744-019-0155-5. Epub 2019 Jun 1. PMID 31154634
- [Derived] Coates LC, Orbai AM, Morita A, Benichou O, Kerr L, Adams DH, Shuler CL, Birt J, Helliwell PS. Achieving minimal disease activity in psoriatic arthritis predicts meaningful improvements in patients' health-related quality of life and productivity. BMC Rheumatol. 2018 Aug 13;2:24. doi: 10.1186/s41927-018-0030-y. eCollection 2018. PMID 30886974
- [Derived] Gladman DD, Orbai AM, Klitz U, Wei JC, Gallo G, Birt J, Rathmann S, Shrom D, Marzo-Ortega H. Ixekizumab and complete resolution of enthesitis and dactylitis: integrated analysis of two phase 3 randomized trials in psoriatic arthritis. Arthritis Res Ther. 2019 Jan 29;21(1):38. doi: 10.1186/s13075-019-1831-0. PMID 30696483
- [Derived] Genovese MC, Combe B, Kremer JM, Tsai TF, Behrens F, Adams DH, Lee C, Kerr L, Nash P. Safety and efficacy of ixekizumab in patients with PsA and previous inadequate response to TNF inhibitors: week 52 results from SPIRIT-P2. Rheumatology (Oxford). 2018 Nov 1;57(11):2001-2011. doi: 10.1093/rheumatology/key182. PMID 30053162
- [Derived] Nash P, Kirkham B, Okada M, Rahman P, Combe B, Burmester GR, Adams DH, Kerr L, Lee C, Shuler CL, Genovese M; SPIRIT-P2 Study Group. Ixekizumab for the treatment of patients with active psoriatic arthritis and an inadequate response to tumour necrosis factor inhibitors: results from the 24-week randomised, double-blind, placebo-controlled period of the SPIRIT-P2 phase 3 trial. Lancet. 2017 Jun 10;389(10086):2317-2327. doi: 10.1016/S0140-6736(17)31429-0. Epub 2017 May 24. PMID 28551073
- See also: Click here for more information about this study: A Study of Ixekizumab (LY2439821) in Participants With Active Psoriatic Arthritis — http://www.lillytrialguide.com/EN-us/studies/arthritis/rhbe

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixekizumab 80 mg Q2W (Ixe 80 mg Q2W)- Blinded Treatment Period: Participants received a starting dose of 160 mg of ixekizumab given as 2 subcutaneous (SC) injections at Week 0 followed by 1 SC injection of 80 mg of ixekizumab every 2 Weeks (Q2W) given on Weeks 2, 4, 6, 8, 10, 12,14, 16, 18, 20, 22, and 24.
- Ixekizumab 80 mg Q4W (Ixe 80 mg Q4W)- Blinded Treatment Period: Participants received a starting dose of 160 mg of ixekizumab given as 2 SC injections at Week 0 followed by 1 SC injection of 80 mg of ixekizumab Q4W given on Weeks 4, 8 and 12 alternating with placebo for ixekizumab injections Q4W given on Weeks 2, 6, 10 and 14, 18, and 22.
- Placebo (PBO) - Blinded Treatment Period: Participants received placebo for ixekizumab as 2 SC injections followed by 1 SC injection Q2W given on Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24.
- Ixe 80 mg Q2W - Blinded Treatment Period IR: Week 16 inadequate responders from the placebo treatment group who were re-randomized (1:1) to ixekizumab 80 mg Q2W and IR from ixekizumab 80 mg Q2W who continued on ixekizumab 80 mg Q2W. Participants received rescue therapy while receiving ixekizumab given as 1 injection of 80 mg Q2W given on Weeks 16, 18, 20, 22, and 24.
- Ixe 80 mg Q4W - Blinded Treatment Period IR: Week 16 inadequate responders from the placebo treatment group who were re-randomized (1:1) to ixekizumab 80 mg Q4W and IR from ixekizumab 80 mg Q4W who continued on ixekizumab 80 mg Q4W. Participants received rescue therapy while receiving ixekizumab given as 1 injection of 80 mg Q4W given on Weeks 16 and 20 alternating with placebo for ixekizumab injections Q4W given on Weeks 18 and 22.
- PBO IR / Ixe 80 mg Q2W - Blinded Treatment Period IR: Participants initially randomized to placebo treatment group in the double blind treatment period who were flagged as inadequate responders at week 16 were re-randomized to ixekizumab 80 mg Q2W for the remainder of the current period and following period.
- PBO IR / Ixe 80 mg Q4W - Blinded Treatment Period IR: Participants initially randomized to placebo treatment group in the double blind treatment period who were flagged as inadequate responders at week 16 were re-randomized to ixekizumab 80 mg Q4W for the remainder of the current period and following period.
- Ixe 80 mg Q2W / Ixe 80 mg Q2W - Extended Treatment Period: Participants who were randomized to ixekizumab 80 mg Q2W at week 0 and continued on ixekizumab 80 mg Q2W during the Extension Period.
- Ixe 80 mg Q4W / Ixe 80 mg Q4W - Extended Treatment Period: Participants who were randomized to ixekizumab 80 mg Q4W at week 0 and continued on ixekizumab 80 mg Q4W during the Extension Period.
- Placebo/ Ixe 80 mg Q2W - Extended Treatment Period: Participants who were randomized to placebo at Week 0 then randomized to ixekizumab 80 mg Q2W during the Extension Period.
  Participants who remained on placebo at the completion of the double blind treatment period received the first dose of ixekizumab (160 mg starting dose) at Week 24.
  Participants who were IRs at Week 16 and were re-randomized to ixekizumab at Week 16 received the first dose of ixekizumab (160 mg starting dose) at Week 16.
- Placebo/ Ixe 80 mg Q4W - Extended Treatment Period: Participants who were randomized to placebo at Week 0 then randomized to ixekizumab 80 mg Q4W during the Extension Period.
  Participants who remained on placebo at the completion of the double blind treatment period received the first dose of ixekizumab (160 mg starting dose) at Week 24.
  Participants who were IRs at Week 16 and were re-randomized to ixekizumab at Week 16 received the first dose of ixekizumab (160 mg starting dose) at Week 16.
- Ixe 80 mg Q2W - Post Treatment Follow-Up Period: Participants who received ixekizumab 80 mg Q2W prior to entering the post-treatment follow-up period, who were either completed the study or discontinued the study early entered the post-treatment follow-up period (a 12-24 week period after their last scheduled treatment visit).
- Ixe 80 mg Q4W - Post Treatment Follow-Up Period: Participants who received ixekizumab 80 mg Q4W prior to entering the post-treatment follow-up period, who were either completed the study or discontinued the study early entered the post-treatment follow-up period (a 12-24 week period after their last scheduled treatment visit).
- PBO - Post Treatment Follow-Up Period: Participants who received PBO prior to entering the post-treatment follow-up period, who were either completed the study or discontinued the study early entered the post-treatment follow-up period (a 12-24 week period after their last scheduled treatment visit).
Period: Double Blind Treatment (Week 0-24)
Arm/Group | Ixekizumab 80 mg Q2W (Ixe 80 mg Q2W)- Blinded Treatment Period | Ixekizumab 80 mg Q4W (Ixe 80 mg Q4W)- Blinded Treatment Period | Placebo (PBO) - Blinded Treatment Period | Ixe 80 mg Q2W - Blinded Treatment Period IR | Ixe 80 mg Q4W - Blinded Treatment Period IR | PBO IR / Ixe 80 mg Q2W - Blinded Treatment Period IR | PBO IR / Ixe 80 mg Q4W - Blinded Treatment Period IR | Ixe 80 mg Q2W / Ixe 80 mg Q2W - Extended Treatment Period | Ixe 80 mg Q4W / Ixe 80 mg Q4W - Extended Treatment Period | Placebo/ Ixe 80 mg Q2W - Extended Treatment Period | Placebo/ Ixe 80 mg Q4W - Extended Treatment Period | Ixe 80 mg Q2W - Post Treatment Follow-Up Period | Ixe 80 mg Q4W - Post Treatment Follow-Up Period | PBO - Post Treatment Follow-Up Period
Started | 123 | 122 | 118 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received Atleast One Dose of Study Drug | 123 | 122 | 118 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 109 | 111 | 94 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 14 | 11 | 24 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 2 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Failure To Meet Randomization | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: IR (Week 16-24)
Arm/Group | Ixekizumab 80 mg Q2W (Ixe 80 mg Q2W)- Blinded Treatment Period | Ixekizumab 80 mg Q4W (Ixe 80 mg Q4W)- Blinded Treatment Period | Placebo (PBO) - Blinded Treatment Period | Ixe 80 mg Q2W - Blinded Treatment Period IR | Ixe 80 mg Q4W - Blinded Treatment Period IR | PBO IR / Ixe 80 mg Q2W - Blinded Treatment Period IR | PBO IR / Ixe 80 mg Q4W - Blinded Treatment Period IR | Ixe 80 mg Q2W / Ixe 80 mg Q2W - Extended Treatment Period | Ixe 80 mg Q4W / Ixe 80 mg Q4W - Extended Treatment Period | Placebo/ Ixe 80 mg Q2W - Extended Treatment Period | Placebo/ Ixe 80 mg Q4W - Extended Treatment Period | Ixe 80 mg Q2W - Post Treatment Follow-Up Period | Ixe 80 mg Q4W - Post Treatment Follow-Up Period | PBO - Post Treatment Follow-Up Period
Started | 0 (Only IR participants were included.) | 0 (Only IR participants were included.) | 0 (Only IR participants were included.) | 17 (IR from ixekizumab 80 mg Q2W only.) | 15 (IR from ixekizumab 80 mg Q4W only.) | 16 (IR from placebo who re-randomized (1:1) to ixekizumab 80 mg Q2W.) | 16 (IR from placebo who re-randomized (1:1) to ixekizumab 80 mg Q4W.) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 16 | 15 | 16 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Long-Term Extension Period (Week 24-156)
Arm/Group | Ixekizumab 80 mg Q2W (Ixe 80 mg Q2W)- Blinded Treatment Period | Ixekizumab 80 mg Q4W (Ixe 80 mg Q4W)- Blinded Treatment Period | Placebo (PBO) - Blinded Treatment Period | Ixe 80 mg Q2W - Blinded Treatment Period IR | Ixe 80 mg Q4W - Blinded Treatment Period IR | PBO IR / Ixe 80 mg Q2W - Blinded Treatment Period IR | PBO IR / Ixe 80 mg Q4W - Blinded Treatment Period IR | Ixe 80 mg Q2W / Ixe 80 mg Q2W - Extended Treatment Period | Ixe 80 mg Q4W / Ixe 80 mg Q4W - Extended Treatment Period | Placebo/ Ixe 80 mg Q2W - Extended Treatment Period | Placebo/ Ixe 80 mg Q4W - Extended Treatment Period | Ixe 80 mg Q2W - Post Treatment Follow-Up Period | Ixe 80 mg Q4W - Post Treatment Follow-Up Period | PBO - Post Treatment Follow-Up Period
Started | 0 | 0 | 0 | 0 (Only included combined extension participants.) | 0 (Only included combined extension participants.) | 0 (Only included combined extension participants.) | 0 (Only included combined extension participants.) | 107 (IxeQ2W participants who entered the long-term extension period.) | 111 (IxeQ4W participants who entered the long-term extension period.) | 46 (Placebo/IxeQ2W participants who entered the long-term extension period.) | 46 (Placebo/IxeQ4W participants who entered the long-term extension period.) | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 55 | 70 | 20 | 23 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 52 | 41 | 26 | 23 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 32 | 25 | 19 | 18 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 2 | 2 | 0 | 0 | 0
Not completed — Unknown/Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 1 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Period: Follow-Up Period (Up to 12-24 Weeks)
Arm/Group | Ixekizumab 80 mg Q2W (Ixe 80 mg Q2W)- Blinded Treatment Period | Ixekizumab 80 mg Q4W (Ixe 80 mg Q4W)- Blinded Treatment Period | Placebo (PBO) - Blinded Treatment Period | Ixe 80 mg Q2W - Blinded Treatment Period IR | Ixe 80 mg Q4W - Blinded Treatment Period IR | PBO IR / Ixe 80 mg Q2W - Blinded Treatment Period IR | PBO IR / Ixe 80 mg Q4W - Blinded Treatment Period IR | Ixe 80 mg Q2W / Ixe 80 mg Q2W - Extended Treatment Period | Ixe 80 mg Q4W / Ixe 80 mg Q4W - Extended Treatment Period | Placebo/ Ixe 80 mg Q2W - Extended Treatment Period | Placebo/ Ixe 80 mg Q4W - Extended Treatment Period | Ixe 80 mg Q2W - Post Treatment Follow-Up Period | Ixe 80 mg Q4W - Post Treatment Follow-Up Period | PBO - Post Treatment Follow-Up Period
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (Only included post-treatment follow-up participants.) | 0 (Only included post-treatment follow-up participants.) | 0 (Only included post-treatment follow-up participants.) | 0 (Only included post-treatment follow-up participants.) | 142 (IxeQ2W participants who entered post-treatment follow-up.) | 145 (IxeQ4W participants who entered post-treatment follow-up.) | 17 (PBO participants who entered post-treatment follow-up.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 133 | 137 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Unknown/Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo: Participants received placebo for ixekizumab as 2 SC injections followed by 1 SC injection Q2W given on Weeks 2, 4, 6, 8, 10, 12 and 14. Inadequate responders at Week 16 receive rescue therapy and re-randomized (1:1) to either ixekizumab group, receiving a starting dose of 160 mg at Week 16 given as 2 SC injections followed by 80 mg given as 1 injection according to ixekizumab regimen: Q2W or Q4W (with placebo every other dose). All other participants continue placebo as 1 injection Q2W given on Weeks 16, 18, 20 and 22
- Ixekizumab 80 mg Q4W: Participants received a starting dose of 160 mg of ixekizumab given as 2 SC injections at Week 0 followed by 1 SC injection of 80 mg of ixekizumab Q4W given on Weeks 4, 8 and 12 alternating with placebo for ixekizumab injections Q4W given on Weeks 2, 6, 10 and 14. Inadequate responders at Week 16 receive rescue therapy while continuing ixekizumab given as 1 injection of 80 mg Q4W given on Weeks 16 and 20 alternating with placebo for ixekizumab injections Q4W given on Weeks 18 and 22. All other participants continue 80 mg given as 1 injection Q2W given on Weeks 16 and 20 alternating with placebo for ixekizumab injections Q4W given on Weeks 18 and 22
- Ixekizumab 80 mg Q2W: Participants received a starting dose of 160 mg of ixekizumab given as 2 SC injections at Week 0 followed by 1 SC injection of 80 mg of ixekizumab Q2W given on Weeks 2, 4, 6, 8, 10, 12 and 14. Inadequate responders at Week 16 receive rescue therapy while continuing ixekizumab given as 1 injection of 80 mg Q2W given on Weeks 16, 18, 20 and 22. All other participants continue 80 mg given as 1 injection Q2W given on Weeks 16, 18, 20 and 22
- Total: Total of all reporting groups
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W | Total
Number analyzed (Participants) | 118 | 122 | 123 | 363
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (10.39) | 52.6 (13.57) | 51.7 (11.85) | 51.9 (12.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 59 | 73 | 194
  Male | 56 | 63 | 50 | 169
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 13 | 35
  Not Hispanic or Latino | 106 | 109 | 109 | 324
  Unknown or Not Reported | 1 | 2 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 7 | 7 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 1 | 1 | 1 | 3
  White | 108 | 111 | 113 | 332
  More than one race | 2 | 2 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Czechia | 8 | 4 | 8 | 20
  United States | 60 | 65 | 63 | 188
  Taiwan | 6 | 6 | 7 | 19
  Poland | 5 | 4 | 5 | 14
  Italy | 0 | 0 | 1 | 1
  United Kingdom | 5 | 6 | 5 | 16
  Australia | 2 | 2 | 3 | 7
  France | 6 | 6 | 5 | 17
  Germany | 11 | 13 | 12 | 36
  Spain | 15 | 16 | 14 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20 Index (ACR20)
Description: ACR20 response is defined as a greater than or equal to (≥) 20% improvement from baseline for tender joint count (TJC) and swollen joint count (SJC) and in at least 3 of the following 5 criteria: Participant's assessment of Joint Pain visual analog scale (VAS), Participant's Global Assessment of Disease Activity VAS (PatGA), Physician's Global Assessment of the Disease Activity VAS (PGA), Participant's Assessment of Physical Function using the Health Assessment Questionnaire Disability Index (HAQ-DI), or Acute Phase Reactant as measured by high sensitivity C-reactive protein (hs-CRP).
Time Frame: Week 24
Population: All randomized participants. Non-responder Imputation (NRI) is applied for inadequate responders at Week 16 and participants who had missing data at Week 24 for any reason including discontinuation.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Percentage of Participants | 19.5 | 53.3 | 48.0
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Other; p < 0.001, Regression, Logistic — model includes: treatment, geographic region, and tumor necrosis factor inhibitor (TNFi) experience (inadequate responder to 1 TNFi, inadequate responder to 2 TNFi, or intolerance to a TNFi); 1) uses a Wald's test , 2) Non-responder imputation (NRI) was used to calculate the response rates; Odds Ratio (OR) = 4.74, 95% CI 2-sided [2.65 to 8.48]
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; model includes: treatment, geographic region, and TNFi experience (inadequate responder to 1 TNFi, inadequate responder to 2 TNFi, or intolerance to a TNFi); Test type: Other — 1) uses a Wald's test , 2) Non-responder imputation (NRI) was used to calculate the response rates; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.79, 95% CI 2-sided [2.12 to 6.78]

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: HAQ-DI is a participant reported questionnaire that measures disease-associated disability(physical function).It consists of 24 questions with 8 domains: dressing/grooming,arising,eating,walking,hygiene,reach,grip and other daily activities. The disability section scores the participant's self-perception on degree of difficulty (0=without any difficulty,1=with some difficulty,2=with much difficulty,3=unable to do)covering the 8 domains.The HAQ-DI is a composite ranging from 0-3 with lower scores indicating less functional disability.The reported use of special aids/devices and/or the need for assistance of another person to perform these activities is assessed.Least Square (LS) mean calculated using Mixed Model Repeated Measurements (MMRM) analysis with treatment,baseline score,geographic region, TNFi experience,visit, treatment-by-visit interaction(itcn), geographic region-by-visit itcn,TNFi experience-by-visit itcn and baseline score-by-visit itcn.
Time Frame: Baseline, Week 24
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
units on a scale | -0.2 (0.08) | -0.6 (0.07) | -0.4 (0.07)

3. Secondary Outcome: Percentage of Participants Achieving ACR20
Description: ACR20 response is defined as a ≥20% improvement from baseline for TJC and SJC and in at least 3 of the following 5 criteria: Participant's assessment of Joint Pain VAS, Participant's Global Assessment of Disease Activity VAS, Physician's Global Assessment of the Disease Activity VAS, Participant's Assessment of Physical Function using the HAQ-DI, or hs-CRP.
Time Frame: Week 12
Population: All randomized participants. NRI is applied for inadequate responders at Week 16 and participants who had missing data at Week 24 for any reason including discontinuation.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Percentage of Participants | 22.0 | 50.0 | 48.0

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50 Index (ACR50)
Description: ACR50 response is defined as a ≥50% improvement from baseline for TJC and SJC and in at least 3 of the following 5 criteria: Participant's assessment of Joint Pain VAS, Participant's Global Assessment of Disease Activity VAS, Physician's Global Assessment of the Disease Activity VAS, Participant's Assessment of Physical Function using the HAQ-DI, or hs-CRP.
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Percentage of Participants | 5.1 | 35.2 | 33.3

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70 Index (ACR70)
Description: ACR70 response is defined as a ≥70% improvement from baseline for TJC and SJC and in at least 3 of the following 5 criteria: Participant's assessment of Joint Pain VAS, Participant's Global Assessment of Disease Activity VAS, Physician's Global Assessment of the Disease Activity VAS, Participant's Assessment of Physical Function using the HAQ-DI, or hs-CRP.
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Percentage of Participants | 0 | 22.1 | 12.2

6. Secondary Outcome: Percentage of Participants With Psoriasis Area and Severity Index (PASI) 75
Description: The PASI is an index that combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation, erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease. Participants achieving PASI 75 were defined as having an improvement of at least 75% in the PASI compared to their baseline measures.
Time Frame: Week 12
Population: All randomized participants with baseline psoriatic lesion(s) involving ≥3% body surface area (BSA). NRI is applied for inadequate responders at Week 16 and participants who had missing data at Week 24 for any reason including discontinuation.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 67 | 68 | 68
Percentage of Participants | 10.4 | 57.4 | 61.8

7. Secondary Outcome: Percentage of Patients Achieving Minimal Disease Activity (MDA)
Description: It uses a composite of 7 key outcome measures (includes PASI) used in PsA to encompass all of the domains of the disease to measure the overall state of a patients' disease. The LEI is used to assess tender entheseal points. Patients are classified as achieving MDA if they fulfill 5 of 7 outcome measures: 1. TJC ≤1, 2. SJC ≤1, 3. PASI total score ≤1 or BSA ≤3, 4. patient pain VAS score of ≤15, 5. patient global VAS score of ≤20, 6. HAQ-DI score ≤0.5, 7. tender entheseal points (6 entheseal points) ≤1.
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Percentage of Participants | 3.4 | 27.9 | 23.6

8. Secondary Outcome: Percentage of Patients Achieving Complete Resolution in Enthesitis as Assessed by the Leeds Enthesitis Index (LEI)
Description: The LEI was developed specifically for use in PsA. It measures enthesitis at 6 sites (lateral epicondyle, left and right; medial femoral condyle, left and right; Achilles tendon insertion, left and right). Each site was assigned a score of 0 (absent) or 1 (present); the results from each site were then added to produce a total score (range 0 to 6). So, "0" indicates good score here.
Time Frame: Week 24
Population: All randomized participants who had baseline enthesitis, baseline LEI score and post baseline LEI score data. NRI is applied for inadequate responders at Week 16 and participants who had missing data at Week 24 for any reason including discontinuation.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 69 | 68 | 84
Percentage of Participants | 21.7 | 35.3 | 31.0

9. Secondary Outcome: Change From Baseline in Itch Numeric Rating Scale (NRS)
Description: The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participants itching from psoriasis was indicated by circling the number that best described the worst level of itching in the past 24 hours. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, TNFi experience, visit, treatment-by-visit interaction, geographic region-by-visit interaction, TNFi experience-by-visit interaction, and baseline score-by-visit interaction.
Time Frame: Baseline, Week 12
Population: All randomized participants who had baseline psoriatic lesion(s) involving >=3% BSA, baseline itch NRS score and post baseline itch NRS score data.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Units on a Scale | -0.7 (0.40) | -3.4 (0.39) | -3.3 (0.39)

10. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC)
Description: TJC is the number of tender and painful joints determined for each participant by examination of 68 joints. Joints were assessed by pressure and joint manipulation on physical examination. Participants were asked for pain sensations on these manipulations and watched for spontaneous pain reactions. Any positive response on pressure, movement, or both was translated into a single tender-versus-nontender dichotomy. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, TNFi experience, visit, treatment-by-visit interaction, geographic region-by-visit interaction, TNFi experience-by-visit interaction, and baseline score-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants with baseline and post baseline TJC data.
Measure: Least Squares Mean (Standard Error); unit: Tender Joint Count
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Tender Joint Count | -6.2 (1.96) | -12.7 (1.87) | -12.5 (1.77)

11. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC)
Description: SJC is the number of swollen joints determined for each participant by examination of 66 joints. Joints were classified as either swollen or not swollen. Swelling was defined as palpable fluctuating synovitis of the joint. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, TNFi experience, visit, treatment-by-visit interaction, geographic region-by-visit interaction, TNFi experience-by-visit interaction, and baseline score-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants with baseline and post baseline SJC data.
Measure: Least Squares Mean (Standard Error); unit: Swollen Joint Count
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Swollen Joint Count | -5.0 (1.05) | -8.5 (0.99) | -7.4 (0.94)

12. Secondary Outcome: Change From Baseline in Participants Assessment of Pain Visual Analog Scale (VAS)
Description: The pain VAS is a participant-administered single-item scale designed to measure current joint pain from Psoriatic arthritis (PsA) using a 100-millimeter(mm) horizontal VAS. Overall severity of participant's joint pain from PsA is indicated by marking a vertical tick on the horizontal 100-mm scale, where the left end from 0 mm (no pain) to right end 100 mm (worst possible joint pain). LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, TNFi experience, visit, treatment-by-visit interaction, geographic region-by-visit interaction, TNFi experience-by-visit interaction, and baseline score-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants with baseline and post baseline TJC and SJC data.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Units on a Scale | -21.4 (3.97) | -36.9 (3.74) | -33.5 (3.58)

13. Secondary Outcome: Change From Baseline in Patients Global Assessment of Disease Activity VAS
Description: The patient's overall assessment of his or her PsA activity will be recorded using a 100-mm horizontal VAS, where 0 represents no disease activity and 100 represents extremely active disease. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, TNFi experience, visit, treatment-by-visit interaction, geographic region-by-visit interaction, TNFi experience-by-visit interaction, and baseline score-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants with baseline and post baseline Patients Global Assessment of Disease Activity VAS score.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Units on a Scale | -19.0 (3.91) | -40.7 (3.68) | -37.3 (3.53)

14. Secondary Outcome: Change From Baseline in Physicians Global Assessment of Disease Activity VAS
Description: The investigator will be asked to give an overall assessment of the severity of the participant's current PsA activity using a 100-mm horizontal VAS, where 0 represents no disease activity and 100 represents extremely active disease. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, TNFi experience, visit, treatment-by-visit interaction, geographic region-by-visit interaction, TNFi experience-by-visit interaction, and baseline score-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants with baseline and post baseline Physicians Global Assessment of Disease Activity VAS score.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Units on a Scale | -18.3 (3.98) | -40.0 (3.85) | -37.9 (3.75)

15. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP)
Description: C-reactive protein (CRP) is a disease related biomarker and measured in milligrams per liter. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, TNFi experience, visit, treatment-by-visit interaction, geographic region-by-visit interaction, TNFi experience-by-visit interaction, and baseline score-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants with baseline and post baseline CRP data.
Measure: Least Squares Mean (Standard Error); unit: milligram per liter (mg/L)
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
milligram per liter (mg/L) | -3.6 (1.87) | -11.8 (1.76) | -9.8 (1.68)

16. Secondary Outcome: Change From Baseline in Disease Activity Score-CRP (DAS28-CRP)
Description: The DAS28-CRP is a measure of disease activity in 28 joints that consists of a composite numerical score with the following variables: TJC28, SJC28, hs-CRP (measured in mg/L), and Participant's Global Assessment of Disease Activity recorded by participants on a 0 to 100 millimeter (mm) VAS. For DAS28-CRP, the Tender Joint Count 28 (TJC28) and Swollen Joint Count (SJC28) are a subset of TJC and SJC, and include 14 joints on each side of the body: 2 shoulders, 2 elbows, 2 wrists, 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees. DAS28 values range from 0 to 9.4. Higher values indicate more severe symptoms and greater functional impairment. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, TNFi experience, visit, treatment-by-visit interaction, geographic region-by-visit interaction, TNFi experience-by-visit interaction, and baseline score-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline and post baseline DAS28-CRP data.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Units on a Scale | -0.8 (0.20) | -2.1 (0.19) | -1.8 (0.18)

17. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score
Description: The BASDAI is a self-administered measure used to answer 6 questions with a 0 to 10 centimeter (cm) VAS pertaining to the 5 major symptoms of axial activity. To give each symptom equal weighting, the mean of the 2 scores relating to morning stiffness was taken. The resulting 0 to 50 score was divided by 5 to give a final 0 to 10 BASDAI Score. BASDAI ranges from 0-10. Higher scores represent greater disease activity. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, TNFi experience, visit, treatment-by-visit interaction, geographic region-by-visit interaction, TNFi experience-by-visit interaction, and baseline score-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline axial involvement defined as baseline BASDAI score >4, baseline BASDAI score and post baseline BASDAI score data.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Units on a Scale | -2.1 (0.38) | -3.7 (0.36) | -3.6 (0.35)

18. Secondary Outcome: Change From Baseline in Fatigue Severity Numeric Rating Scale (NRS) Score
Description: The Fatigue Severity NRS is a participant-administered single-item 11-point horizontal scale anchored at 0 and 10, with 0 representing "no fatigue" and 10 representing "as bad as you can imagine." Participants rated their fatigue (feeling tired or worn out) by circling the 1 number that described their worst level of fatigue during the past 24 hours. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, TNFi experience, visit, treatment-by-visit interaction, geographic region-by-visit interaction, TNFi experience-by-visit interaction, and baseline score-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline and post baseline fatigue NRS data.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Units on a Scale | -0.7 (0.37) | -2.0 (0.35) | -2.1 (0.34)

19. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Scores: Physical Component Summary (PCS)
Description: The SF-36 is a participant-reported outcome measure evaluating participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. The 8 domains are regrouped into the PCS and MCS scores. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health. In this study, the SF-36 acute version was used, which has a 1 week recall period. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, TNFi experience, visit, treatment-by-visit interaction, geographic region-by-visit interaction, TNFi experience-by-visit interaction, and baseline score-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline and post baseline PCS data.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Units on a Scale | 3.3 (1.36) | 8.9 (1.29) | 8.2 (1.23)

20. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Scores: Mental Component Summary (MCS)
Description: as for outcome 19
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline and post baseline MCS data.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 118 | 122 | 123
Units on a Scale | 0.9 (1.32) | 3.6 (1.24) | 4.0 (1.18)

21. Secondary Outcome: Number of Participants With Treatment Emergent Anti-Drug Antibodies (TE-ADA)
Description: Number of participants with positive treatment emergent anti-ixekizumab antibodies was summarized by treatment group.
Time Frame: Week 24
Population: All randomized participants who received at least 1 dose of ixekizumab and had evaluable anti-ixekizumab antibody measurement.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 112 | 117 | 120
Participants | 1 | 8 | 4

22. Secondary Outcome: Pharmacokinetics (PK):Minimum Observed Serum Concentration at Steady State (Ctrough,ss) of Ixekizumab
Description: The Ctrough is the minimum observed serum concentration at steady state of Ixekizumab. The Ctrough at Week 24 was reported.
Time Frame: All immunogenicity samples post the first Ixekizumab dose (Week 4, 12, 24, 36, and 52) and PK samples collected per dedicated sparse sampling plan (4-5 samples per patient) across Weeks 1 through 24 and Early termination visit (ETV)
Population: The PK Population included all enrolled participants who received at least one dose of the study drug and had evaluable ixekizumab PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micograms per milliliter (mcg/mL)
Arm/Group | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 102 | 101
micograms per milliliter (mcg/mL) | 2.46 (79.1) | 7.96 (71.1)

23. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve for Dosing Interval (Tau) at Steady State [AUC(Tau,Steady State)] of Ixekizumab
Description: The AUC(Tau,Steady State) is the area under the concentration-time curve for dosing interval (Tau) at steady state of ixekizumab (Tau is 28 days for 80 mg Q4W cohort, and is 14 days for 80mg Q2W cohort, respectively).
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*day/mL
Arm/Group | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 100
mcg*day/mL | 141 (59.3) | 143 (57.5)

24. Secondary Outcome: Percentage of Participants Achieving ACR 20
Description: as for outcome 3
Time Frame: Week 52 and Week 156
Population: All randomized participants. Non-responder Imputation (NRI) is applied for inadequate responders at week 16 and participants who discontinued on or prior to week 24.
Measure: Number; unit: Percentage of participants
Arm/Group | Ixe 80 mg Q2W / Ixe 80 mg Q2W - Extended Treatment Period | Ixe 80 mg Q4W / Ixe 80 mg Q4W - Extended Treatment Period | Placebo/ Ixe 80 mg Q2W - Extended Treatment Period | Placebo/ Ixe 80 mg Q4W - Extended Treatment Period
Number analyzed (Participants) | 107 | 111 | 46 | 46
Percentage of participants
  Week 52 | 58.9 | 67.6 | 50.0 | 60.9
  Week 156 | 42.1 | 50.5 | 39.1 | 45.7

25. Secondary Outcome: Percentage of Participants Achieving ACR 50
Description: as for outcome 4
Time Frame: Week 52 and Week 156
Population: as for outcome 24
Measure: Number; unit: Percentage of participants
Arm/Group | Ixe 80 mg Q2W / Ixe 80 mg Q2W - Extended Treatment Period | Ixe 80 mg Q4W / Ixe 80 mg Q4W - Extended Treatment Period | Placebo/ Ixe 80 mg Q2W - Extended Treatment Period | Placebo/ Ixe 80 mg Q4W - Extended Treatment Period
Number analyzed (Participants) | 107 | 111 | 46 | 46
Percentage of participants
  Week 52 | 38.3 | 45.9 | 34.8 | 43.5
  Week 156 | 29.0 | 35.1 | 26.1 | 34.8

26. Secondary Outcome: Percentage of Participants Achieving ACR 70
Description: as for outcome 5
Time Frame: Week 52 and Week 156
Population: as for outcome 24
Measure: Number; unit: Percentage of participants
Arm/Group | Ixe 80 mg Q2W / Ixe 80 mg Q2W - Extended Treatment Period | Ixe 80 mg Q4W / Ixe 80 mg Q4W - Extended Treatment Period | Placebo/ Ixe 80 mg Q2W - Extended Treatment Period | Placebo/ Ixe 80 mg Q4W - Extended Treatment Period
Number analyzed (Participants) | 107 | 111 | 46 | 46
Percentage of participants
  Week 52 | 20.6 | 28.8 | 15.2 | 23.9
  Week 156 | 22.4 | 21.6 | 10.9 | 19.6

ADVERSE EVENTS:
Time Frame: Baseline Up To 2.55 Years
Description: All randomized participants who received at least one dose of study drug. The gender specific events only occurring in male or female participants were adjusted accordingly.
Groups:
- Ixe 80 mg Q2W - Blinded Treatment Period IR: Week 16 inadequate responders from the placebo treatment group who were re-randomized (1:1) to ixekizumab 80 mg Q2W and IR from ixekizumab 80 mg Q2W who continued on ixekizumab 80 mg Q2W. Patients receive rescue therapy while receiving ixekizumab given as 1 injection of 80 mg Q2W given on Weeks 16, 18, 20, 22, and 24.
- Ixe 80 mg Q4W - Blinded Treatment Period IR: Week 16 inadequate responders from the placebo treatment group who were re-randomized (1:1) to ixekizumab 80 mg Q4W and IR from ixekizumab 80 mg Q4W who continued on ixekizumab 80 mg Q4W. Patients receive rescue therapy while receiving ixekizumab given as 1 injection of 80 mg Q4W given on Weeks 16 and 20 alternating with placebo for ixekizumab injections Q4W given on Weeks 18 and 22.
- PBO IR / Ixe 80 mg Q2W - Blinded Treatment Period IR: Participants initially randomized to placebo treatment group in the double blind treatment period who were flagged as inadequate responders as week 16 were re-randomized to ixekizumab 80 mg Q2W for the remainder of the current period and following period.
- PBO IR / Ixe 80 mg Q4W - Blinded Treatment Period IR: Participants initially randomized to placebo treatment group in the double blind treatment period who were flagged as inadequate responders as week 16 were re-randomized to ixekizumab 80 mg Q4W for the remainder of the current period and following period.
Arm/Group | Ixekizumab 80 mg Q2W (Ixe 80 mg Q2W)- Blinded Treatment Period | Ixekizumab 80 mg Q4W (Ixe 80 mg Q4W)- Blinded Treatment Period | Placebo (PBO) - Blinded Treatment Period | Ixe 80 mg Q2W - Blinded Treatment Period IR | Ixe 80 mg Q4W - Blinded Treatment Period IR | PBO IR / Ixe 80 mg Q2W - Blinded Treatment Period IR | PBO IR / Ixe 80 mg Q4W - Blinded Treatment Period IR | Ixe 80 mg Q2W / Ixe 80 mg Q2W - Extended Treatment Period | Ixe 80 mg Q4W / Ixe 80 mg Q4W - Extended Treatment Period | Placebo/ Ixe 80 mg Q2W - Extended Treatment Period | Placebo/ Ixe 80 mg Q4W - Extended Treatment Period | Ixe 80 mg Q2W - Post Treatment Follow-Up Period | Ixe 80 mg Q4W - Post Treatment Follow-Up Period | PBO - Post Treatment Follow-Up Period
Serious Adverse Events (participants affected / at risk) | 8/123 | 3/122 | 4/118 | 0/17 | 0/15 | 0/16 | 1/16 | 10/107 | 13/111 | 6/46 | 3/46 | 1/142 | 2/145 | 2/17
Other Adverse Events (participants affected / at risk) | 58/123 | 58/122 | 40/118 | 5/17 | 8/15 | 11/16 | 8/16 | 59/107 | 65/111 | 20/46 | 32/46 | 16/142 | 13/145 | 2/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ixekizumab 80 mg Q2W (Ixe 80 mg Q2W)- Blinded Treatment Period (N=123) | Ixekizumab 80 mg Q4W (Ixe 80 mg Q4W)- Blinded Treatment Period (N=122) | Placebo (PBO) - Blinded Treatment Period (N=118) | Ixe 80 mg Q2W - Blinded Treatment Period IR (N=17) | Ixe 80 mg Q4W - Blinded Treatment Period IR (N=15) | PBO IR / Ixe 80 mg Q2W - Blinded Treatment Period IR (N=16) | PBO IR / Ixe 80 mg Q4W - Blinded Treatment Period IR (N=16) | Ixe 80 mg Q2W / Ixe 80 mg Q2W - Extended Treatment Period (N=107) | Ixe 80 mg Q4W / Ixe 80 mg Q4W - Extended Treatment Period (N=111) | Placebo/ Ixe 80 mg Q2W - Extended Treatment Period (N=46) | Placebo/ Ixe 80 mg Q4W - Extended Treatment Period (N=46) | Ixe 80 mg Q2W - Post Treatment Follow-Up Period (N=142) | Ixe 80 mg Q4W - Post Treatment Follow-Up Period (N=145) | PBO - Post Treatment Follow-Up Period (N=17)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basedow's disease (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Latent tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/50 (0) | 1/63 (1) | 0/56 (0) | 0/5 (0) | 0/9 (0) | 0/10 (0) | 0/9 (0) | 0/46 (0) | 0/56 (0) | 0/24 (0) | 0/20 (0) | 0/64 (0) | 0/72 (0) | 0/9 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/73 (1) | 0/59 (0) | 0/62 (0) | 0/12 (0) | 0/6 (0) | 0/6 (0) | 0/7 (0) | 0/61 (0) | 0/55 (0) | 0/22 (0) | 0/26 (0) | 0/78 (0) | 0/73 (0) | 0/8 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adnexa uteri cyst (Reproductive system and breast disorders) | 0/73 (0) | 0/59 (0) | 1/62 (1) | 0/12 (0) | 0/6 (0) | 0/6 (0) | 0/7 (0) | 0/61 (0) | 0/55 (0) | 0/22 (0) | 0/26 (0) | 0/78 (0) | 0/73 (0) | 0/8 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1/73 (1) | 0/59 (0) | 0/62 (0) | 0/12 (0) | 0/6 (0) | 0/6 (0) | 0/7 (0) | 0/61 (0) | 0/55 (0) | 0/22 (0) | 0/26 (0) | 0/78 (0) | 0/73 (0) | 0/8 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ixekizumab 80 mg Q2W (Ixe 80 mg Q2W)- Blinded Treatment Period (N=123) | Ixekizumab 80 mg Q4W (Ixe 80 mg Q4W)- Blinded Treatment Period (N=122) | Placebo (PBO) - Blinded Treatment Period (N=118) | Ixe 80 mg Q2W - Blinded Treatment Period IR (N=17) | Ixe 80 mg Q4W - Blinded Treatment Period IR (N=15) | PBO IR / Ixe 80 mg Q2W - Blinded Treatment Period IR (N=16) | PBO IR / Ixe 80 mg Q4W - Blinded Treatment Period IR (N=16) | Ixe 80 mg Q2W / Ixe 80 mg Q2W - Extended Treatment Period (N=107) | Ixe 80 mg Q4W / Ixe 80 mg Q4W - Extended Treatment Period (N=111) | Placebo/ Ixe 80 mg Q2W - Extended Treatment Period (N=46) | Placebo/ Ixe 80 mg Q4W - Extended Treatment Period (N=46) | Ixe 80 mg Q2W - Post Treatment Follow-Up Period (N=142) | Ixe 80 mg Q4W - Post Treatment Follow-Up Period (N=145) | PBO - Post Treatment Follow-Up Period (N=17)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Entropion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 4 (20) | 3 (4) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (6) | 1 (1) | 2 (4) | 2 (4) | 0 (0) | 1 (3) | 0 (0) | 3 (7) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 15 (47) | 6 (20) | 1 (1) | 2 (3) | 1 (2) | 2 (2) | 1 (2) | 6 (92) | 2 (39) | 4 (7) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 2 (15) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (46) | 1 (1) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 1 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 11 (12) | 11 (13) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 9 (11) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 15 (26) | 20 (32) | 6 (11) | 4 (6) | 3 (4) | 5 (5) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 5 (7) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 10 (14) | 11 (13) | 4 (4) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (4) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 12 (12) | 12 (14) | 9 (12) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 20 (33) | 15 (23) | 4 (7) | 8 (9) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 6 (11) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (13) | 7 (8) | 1 (1) | 5 (9) | 2 (3) | 0 (0) | 2 (2)
Vulvovaginal candidiasis (Infections and infestations) | 2/73 (2) | 0/59 (0) | 0/62 (0) | 1/12 (1) | 0/6 (0) | 0/6 (0) | 0/7 (0) | 0/61 (0) | 1/55 (1) | 0/22 (0) | 1/26 (1) | 0/78 (0) | 0/73 (0) | 0/8 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 2/73 (2) | 1/59 (1) | 1/62 (1) | 0/12 (0) | 0/6 (0) | 0/6 (0) | 0/7 (0) | 2/61 (2) | 0/55 (0) | 0/22 (0) | 2/26 (2) | 0/78 (0) | 0/73 (0) | 0/8 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 8 (9) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 1 (1) | 1 (1) | 1 (4) | 1 (1) | 6 (6) | 0 (0)
Sleep terror (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/50 (1) | 0/63 (0) | 0/56 (0) | 0/5 (0) | 0/9 (0) | 0/10 (0) | 0/9 (0) | 1/46 (1) | 1/56 (1) | 1/24 (1) | 3/20 (3) | 0/64 (0) | 0/72 (0) | 0/9 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (5) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 6 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days